CLINICAL TRIAL: NCT03678376
Title: Identification of Neurocognitive Disorders by General Practitioners in Primary Care
Acronym: TROCOMEGE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL18_0041
Record Dates: First submitted 2018-09-11; First posted 2018-09-19 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Neurocognitive Disorders
Keywords: Diagnostic strategy; Neurocognitive disorders; Primary Care
MeSH Terms: conditions — Neurocognitive Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- complaint, cognitive and functional assessments (Other): All patients will be included in a single arm. They will complete an evaluation with their General Practitioner, followed by an evaluation at the Memory Clinic with a specialist (neurologist, geriatrician or psychiatrist).
  Interventions: Other: complaint, cognitive and functional assessments

INTERVENTIONS:
Other: complaint, cognitive and functional assessments — The evaluation with their GP is composed of (1-) Clinical impression, (2-) GP-Cog part 2 with patient or their informal caregiver and (3-) 6-CIT test.
  The identification of patients at risk of NCD with the new strategy applied by the GP will be compared to the gold standard for diagnosis of NCD at the Memory Clinic, established according to Diagnosis and Statistical Manual of mental disorders (DSM-5) criteria and based on a clinical, neuropsychological evaluation and functional abilities. If needed, a secondary etiological diagnosis procedure will be undertaken following the HAS 2011 recommendation including brain MRI and biology.
  Other Names: Evaluation of a new rapid diagnostic strategy for general practitioners assessing complaint, cognition and autonomy in primary care to identify neurocognitive disorders at different stages

SUMMARY:
Neurocognitive disorders (NCD) are today often largely underdiagnosed or diagnosed in late stages in France. Indeed the ALzheimer COoperative Valuation in Europe (ALCOVE) study stated that about 50% of people living with NCD remain undiagnosed until late severe stages with a deep autonomy loss inducing at risk behaviours and/or behavioural crisis. The French High Authority of Health (Haute Autorité de Santé - HAS) and ALCOVE recommend a timely diagnosis at a time when the specific intervention help to implement secondary or tertiary prevention dynamics that would delay severe complications and help to maintain a reasonable quality of life for both the patient and the caregiver. Moreover, the representatives of the National College of General Practitioners, the French Federation of Memory Centres, the French Federation of Gerontology and Geriatrics, the French Federation of Neurology, the French Society of Psychogeriatrics and the National Plan on Neurodegenerative Diseases designed a hierarchized and tailored diagnosis strategy of NCD promoting a shared diagnosis between the General Practitioner (GP) and specialists of NCD. It therefore appears crucial to determine the diagnosis value of a short duration strategy assessing the complaint, cognition and autonomy in primary care to detect NCD and referring to a specialist to perform the etiological diagnosis. The identification of NCD by GP in primary care (TROCOMEGE) study aims at assessing the positive and negative predictive values of a NCD diagnosis strategy through the assessment of the subjective memory complaint, the cognitive status and the autonomy level in primary care. It relies on the clinical impression of the GP, a cognitive complaint interview for complaint and functional assessment thanks to the General Practitioner assessment of Cognition (GP-Cog, part 2) tool and the cognitive assessment thanks to the Six-Item Cognitive Impairment test (6-CIT).

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 65 and over,
* Patient expressing a cognitive complaint (memory, language, sense of time and place disorientation for example) to his/her general practitioner; the complaint can be provided by an informal caregiver and /or, presenting with "at risk" behaviour* possibly related to a NCD (mistaking medicine or forgetting medical consultation, forgetting hot meals, losing him/herself for example…),
* Patients able to understand the specifications of the study and to realize it (vision, audition, language…)
* Patient who has been informed and has consented to the study (himself/herself and by a trusted person/a family member if applicable) as established by the "article L. 1121-8 du Code de la Santé Publique".
* Registered with a social security system

Exclusion Criteria:

* Institutionalized patients
* Patients unable to understand the purpose of the study,
* Patients with neurocognitive disorders already diagnosed
* Patients under legal protection
* Patients with auditory or visual disorders which do not allow to perform the assessment
* Patients who do not want to go to the Memory Clinic
* Patients with severe disease commit the prognosis in relatively short term
* Participation to another trial that would interfere with the present study
* Patient with severe anxiety or depression preventing from any reliable neuropsychological assessment.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1018 (Estimated)
Dates: Start 2020-02-17 (Actual); Primary Completion 2024-08-17 (Estimated); Study Completion 2024-08-17 (Estimated)

PRIMARY OUTCOMES:
NCD diagnosis established by the GP by clinical impresson | At inclusion
  the GP will have to respond to the following issues 1- Does he think the patient presents a suspect cognitive complaint (Yes/No) 2- does he think the patient presents with a NCD (Yes/No),
NCD diagnosis established by the GP using the GP-Cog part 2 | At inclusion
  * a GP-cog score of 0-3 means no significant cognitive impairment
  * a GP-cog score of 4-6 means significant cognitive complaint
NCD diagnosis established by the GP using the 6-CIT test | At inclusion
  * a 6-CIT score between 0 and 7 means normal, referral not indicated at present
  * a 6-CIT score between 8 and 28 means mild or significant cognitive impairment
NCD diagnosis established in the memory clinics as reference by the Neuropsychologist using the DSM-5 | at 3 months

SECONDARY OUTCOMES:
minor or major NCD diagnosis established by the GP | At inclusion
minor or major NCD diagnosis established by the neuropsychologist using the DSM-5 | At 3 months
diagnosis value of each components of the GP strategy solely or in combination | At inclusion
  Sensitivity, Specificity, Positive Predictive Value, Negative Predictive Value, likelihood ratios will be calculated.
level of cognitive performance established with the Mini Mental State Examination (MMSE) | At 3 months
  A MMSE<18 being is considered as abnormal, MMSE between 18-23 is considered as questionable and MMSE >=24 is considered as normal)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Krolak Salmon, Pr, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital des Charpennes, Villeurbanne, France